CLINICAL TRIAL: NCT04798612
Title: Effect of Low-dose Interferon-alfa2a on Peri-operative Immune Suppression
Acronym: IPOS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJ-874
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — peginterferon alfa-2a; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blinded placebo-controlled phase 2 study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Two 45 mikrogram doses of interferon-alfa2a (Pegasys). Both will be applied subcutanously. First dose is at least one week before surgery. Second dose on the day of surgery before the procedure.
  Interventions: Drug: Pegasys
- Placebo (Placebo Comparator): Two 1 ml doses of saline liquid. Both will be applied subcutanously. First dose is at least one week before surgery. Second dose on the day of surgery before the procedure.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Pegasys — 45 mikrograms of Pegasys. Two subcutanous doses will be administered with at least 7 days in between
  Arms: Intervention arm
Drug: Saline — 0.50 ml of Saline. Two subcutanous doses will be administered with at least 7 days in between
  Arms: Placebo

SUMMARY:
The aim of this randomized double-blinded placebo-controlled phase 2 study is to determine efficacy of preoperative treatment with interferon-alfa2a in patients with pMMR colon cancer on perioperative immune suppression and infiltration of lymphocytes in the primary tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age.
* Patients diagnosed with pMMR colonic adenocarcinoma and scheduled for laparoscopic hemicolectomy.
* ASA class I-III (Classification of the American Society of Anesthesiology)

Exclusion Criteria:

* Patients with childbearing potential without a negative pregnancy test before initiating study drug and / or non-acceptance to the use of contraceptive methods *
* ECOG score function> / = 3
* Current liver or renal disease.
* Severe heart disease
* Previous depression diagnosed by a psychiatrist or in treatment with antidepressant
* Autoimmune disease.
* Uncontrolled thyroid disease.
* Patients who are or have recently (within 6 months) received treatment with immunosuppressive agents other than corticosteroid treatment.
* Epilepsy and / or other serious CNS disorders.
* Patients that have undergone major surgery within one month before planned colon resection.
* Known hypersensitivity to recombinant interferon or auxiliary products of Pegasys®.

  * Spiral, pill, implant, transdermal patch, vaginal ring or depot injection. Sterile / infertile subjects are exempt from the use of contraception. To be considered sterile or infertile must generally be surgical sterilization (vasectomy, bilateral tubectomy, hysterectomy or ovariectomy) or be postmenopausal, defined as absent menstruation for at least 12 months prior to study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Flow-analysis of lymphocytic subpopulations in blood | Change between day of surgery (day 7-14 after first treatment) and postoperative day 1.
  Change in CD3, CD4, and CD8 between intervention and placebo groups
T-cell infiltration in tumor | Day of surgery (day 7-14 after first treatment)
  Difference in CD3, CD4 and CD8 T-cell infiltration between intervention and placebo groups

SECONDARY OUTCOMES:
Quality of recovery (QoR-15) | Third postoperative day and postoperative day 12-16
  Difference in QoR-15 between intervention and placebo groups
Multiplex gene assay - NanoString Pan Cancer 360 IO panel analysis in blood and resected tumor | Day of first treatment (Day 0) and day of surgery (day 7-14 after first treatment)
  Difference in gene expressions between intervention and placebo groups
cfDNA analysis in blood | Day of first treatment (Day 0), day of surgery (day 7-14 after first treatment), postoperative day 2, postoperative day 12-16, and postoperative day 28-32.
  Difference between intervention and placebo groups
Multiplex gene assay - NanoString Pan Cancer 360 IO panel analysis of tumor biopsy and resected specimen | Day of standard endoscopic biopsy (Day -7-14 before treatment) and day of surgery (day 7-14 after first treatment)
  Difference in gene expressions in tumor biopsies and resected specimen between intervention and placebo groups
CRP and neutrophil/lymphocyte ratio | Day of surgery (day 7-14 after first treatment)
  Difference in CRP and neutrophil/lymphocyte ratio between intervention and placebo groups
Immunological and inflammatory cytokines and interleukins | Day of surgery (day 7-14 after first treatment) and postoperative day 1.
  Difference between intervention and placebo groups

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev University Hospital, Herlev, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided